CLINICAL TRIAL: NCT05331495
Title: Prospective Study on the Effect of Intraoperative Hemoperfusion on CIRP Expression and Acute Kidney Injury After Aortic Dissection
Brief Title: Effects of Intraoperative Hemoperfusion on Acute Kidney Injury After Aortic Dissection
Acronym: EIHPOAKIAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2021CRF-029
Record Dates: First submitted 2022-04-10; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-04

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemoperfusion and CPB and DHCA surgery (Experimental): The experimental group was treated with hemoperfusion simultaneously with CPB and DHCA.
  Interventions: Device: Intraoperative Hemoperfusion
- traditional CPB and DHCA surgery (No Intervention): The control group was treated with intraoperative CPB and DHCA surgery.

INTERVENTIONS:
Device: Intraoperative Hemoperfusion — During the operation, the hemoperfusion device and the membrane oxygenator of the extracorporeal circulation device were operated in parallel.
  Arms: Hemoperfusion and CPB and DHCA surgery

SUMMARY:
Acute kidney injury (AKI) is a common and serious complication after aortic dissection (AD), and it is closely related to the inflammatory response associated with cardiopulmonary bypass. Hemoperfusion can reduce the level of systemic inflammatory response effectively in patients with sepsis. Some studies have tried to apply hemoperfusion to cardiopulmonary bypass surgery, and put forward the concept of "absorptive cardiopulmonary bypass", but there are few related research reports. The use of hemoperfusion during cardiopulmonary bypass can reduce the level of systemic inflammatory response, thereby reducing the risk of postoperative AKI and improving the prognosis of patients. The Cardiovascular Surgery Department of the First Affiliated Hospital of Jiaotong University is one of the first demonstration units of "adsorption-type cardiopulmonary bypass" in China. Our previous retrospective analysis shown that intraoperative hemoperfusion can effectively reduce the occurrence of postoperative AKI in patients with AD, compared with traditional cardiopulmonary bypass. In addition, previous studies have found that the increased expression of CIRP after cardiopulmonary bypass can aggravate the oxidative stress and mitochondrial dynamics disorder in renal tubular epithelial cells, thereby inducing AKI. This project is a single-center randomized controlled study. It intends to investigate whether the application of hemoperfusion during cardiopulmonary bypass in patients with AD to reduce the level of systemic inflammatory response can reduce the incidence of postoperative AKI and improve the patient's discharge outcome. At the same time, exploratory studies were conducted to investigate whether hemoperfusion could effectively reduce the expression level of CIRP in the circulation. The successful implementation of this study can provide effective intervention methods and related theoretical basis for reducing the risk of AKI after aortic dissection.

DETAILED DESCRIPTION:
The aim of this study is to explore the effect of hemoperfusion during cardiopulmonary bypass (CPB) on the expression of CIRP in serum after aortic dissection and the incidence of postoperative acute kidney injury (AKI). The subjects of the study are patients with aortic dissection of Stanford type A (AAD) who were treated in the First Affiliated Hospital of Xi'an Jiaotong University and required surgical treatment in cardiovascular surgery. The main types of surgery are ascending aortic replacement or Bentall and Sun's surgery, and all of them undergo deep hypothermic circulatory arrest (DHCA).

The general process of this study is that the patients with AAD treated in our hospital who needed surgical treatment were randomly divided into two groups according to the inclusion and exclusion criteria. The control group was treated with intraoperative CPB and DHCA, and the experimental group was treated with hemoperfusion simultaneously with CPB and DHCA. By detecting the expression level of CIRP in the postoperative serum and the incidence of AKI within 7 days after the operation, the prognosis difference between the two groups was analyzed.

Follow-up content: Collect preoperative clinical data, that is, general information of patients: hospital number, name, gender, age, BMI, smoking history, history of hypertension, diabetes, myocardial infarction and angina pectoris, history of chronic obstructive pulmonary disease, peripheral vascular disease, and brain vascular accident, cardiac function classification, cardiac ultrasonography EF value, preoperative creatinine level, eGFR, cystatin C level, hemoglobin Hct, preoperative CTA results whether the lesion involved renal artery and whether preoperative poor organ perfusion performance. The main evaluation index of postoperative follow-up was whether AKI occurred within 7 days after surgery. The diagnostic criteria for AKI were based on the KDIGO diagnostic criteria. The secondary evaluation criteria were the expression level of serum CIRP 24 hours after surgery, and the changes in the expression level of serum inflammatory factors within 7 days after surgery, and the postoperative survival rate, ventilator assistance time, ICU hospitalization time, postoperative hospitalization time, infection and SOFA score.

The criteria for the termination or withdrawal of the study subjects were that the family members of the patients gave up the follow-up treatment due to personal reasons (economic reasons, etc.), or coronary artery bypass grafting was required due to lesions during the operation, or serious complications such as poor cardiac resuscitation and difficulty in hemostasis occurred or ECMO assistance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 75 years old;
* Patients had aortic dissection type A with onset within 7 days.

Exclusion Criteria:

* Preoperative CTA suggests unilateral or bilateral renal artery false lumen blood supply;
* Past history of renal insufficiency;
* Difficulty in hemostasis during operation due to taking anticoagulant and antiplatelet drugs for various reasons before operation, and the CPB time exceeds 4 hours;
* Severe organ perfusion before surgery, such as lower extremity ischemia or preoperative coma;
* BMI>40 Kg/m^2 or pregnancy status.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | 7 days after surgery
  The serum creatinine of the patients was collected, combined with KDIGO criteria to judge the occurrence and staging of acute kidney injury.

SECONDARY OUTCOMES:
the expression level of serum CIRP | 24 hours after surgery
  The expression level of serum CIRP in patients after operation.
the expression level of serum inflammatory factor | 7 days after surgery
  Changes in the expression levels of serum inflammatory factors within 7 days after surgery;

CONTACTS AND LOCATIONS:
Overall Officials: Xinglong Zheng, PhD, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China